CLINICAL TRIAL: NCT07213076
Title: A Retrospective Study of Treatment Patterns and Clinical Outcomes in Australian EGFR Mutant Advanced and Metastatic Non-Small Cell Lung Cancer NSCLC Patients: First-line and Second-line Osimertinib Usage
Brief Title: Australian Retrospective Analysis of EGFRm Advanced & Metastatic NSCLC Patients Treated With 1L or 2L Osimertinib.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: D5161R00071
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, observational study of treatment patterns and clinical outcomes in Australian EGFRm advanced and metastatic non-small cell lung cancer patients treated with first-line osimertinib or second-line osimertinib.

DETAILED DESCRIPTION:
This study utilizes secondary data collected as part of the AUstralasian thoRacic cancers lOngitudinal cohoRt study and biobAnk (AURORA), which is registered on the Australian New Zealand Clinical Trial Registry: ACTRN12625000038493.

Objectives: In stage IIIB-IV patients with EGFRm NSCLC treated with Osimertinib in the 1L or T790M+ 2L setting in Australia:

Primary Objectives: To describe the Osimertinib Time to Treatment Discontinuation (TTD) in the 1L and 2L settings (as separate cohorts).

Secondary Objectives: To describe the real-world progression-free survival (rwPFS), overall survival (OS), time to next treatment (TTNT) after Osimertinib, patient demographics and clinical characteristics, patterns of care (e.g additional therapies received during and after Osimertinib) in 1L and 2L (T790M+) patients (as separate cohorts).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at least 18 years.
* Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy, patients with relapsed/recurrent disease and prior treatment in early-stage setting allowed.
* The tumour harbours an activating EGFR mutation
* Enrolled in the AURORA registry
* Patients must be either:

  * treatment-naïve for advanced NSCLC (allowing up to 2-cycles of bridging chemotherapy prior to molecular testing results) and initiated 1L Osimertinib per PBS restrictions from August 2020 to December 2022.
  * Previously treated with 1st or 2nd generation EGFR TKIs (gefitinib, erlotinib or afatinib) and confirmed T790M+ EGFRm at disease progression and initiated second-line Osimertinib per PBS restrictions from January 2016 to December 2022.

Exclusion Criteria:

There are no predefined exclusion criteria.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with locally advanced or metastatic NSCLC with an activating EGFR mutation, not amenable to curative surgery or radiotherapy.
  This study consists of two patient cohorts:
  1. L Osimertinib: treatment-naïve for advanced NSCLC and initiated 1L Osimertinib per PBS restrictions.
  2. L (T790M+) Osimertinib: previously treated with 1st or 2nd generation EGFR TKIs, confirmed T790M+ EGFRm at disease progression and initiated 2L Osimertinib per PBS restrictions.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2025-07-04 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Time to Treatment Discontinuation | minimum of 24 months follow up
  up to 5 years follow up for 1L cohort and 9 years follow up for 2 L cohort

SECONDARY OUTCOMES:
rwPFS | minimum 24 months follow up
  up to 5 years follow up for 1L cohort and 9 years follow up for 2L cohort
OS | 12 and 24 months
  up to 5 years follow up for 1L cohort and 9 years follow up for 2L cohort
time to next treatment (TTNT) | minimum 24 months of follow up
  up to 5 years follow up for 1L cohort and 9 years follow up for 2L cohort
baseline demographic and clinical characteristics | at baseline
Details of therapies given concurrently with Osimertinib | up to 1 year post study activation
  up to 5 years follow up for 1L cohort and 9 years follow up for 2L cohort
Details of therapies given subsequent to Osimertinib | up to 1 year post study activation
  up to 5 years follow up for 1L cohort and 9 years follow up for 2L cohort

CONTACTS AND LOCATIONS:
Overall Officials: Marliese Alexander, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Ben Solomon, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Research Site, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data may be requested by researchers, academics, industry, or other individuals/organisations, with each request reviewed for appropriateness on a case-by-case basis by the AURORA Chair and Steering Committee.
  Data sharing requests to be emailed to: AURORA@petermac.org
  Diagnostics, Clinical and Outcomes IPD may be shared.
Supporting Information: Study Protocol
Time Frame: Once the study is complete and reported.
Access Criteria: Each request reviewed for appropriateness on a case-by-case basis by the AURORA Chair and Steering Committee.
URL: https://anzctr.org.au/Trial/Registration/TrialReview.aspx?ACTRN=12625000038493

REFERENCES:
- See also: AURORA ANZCTR registration — https://anzctr.org.au/Trial/Registration/TrialReview.aspx?ACTRN=12625000038493